CLINICAL TRIAL: NCT07148583
Title: Evaluation of the Efficacy and Safety of the Multistrain Probiotic "BioAmicus Complete" in Improving Gastrointestinal Symptoms in Children Aged 0-24 Months: A Randomized, Open-Label, Parallel-Group, Controlled Trial
Brief Title: BioAmicus Complete for Functional Gastrointestinal Symptoms in Infants Aged 0 to 24 Months
Acronym: CTBE2503
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTBE.25.03; Protocol No.: CTBE.25.03 (Other: Clinical Trial and Bioequivalence Center - Hai Phong University of Medicine and Pharmacy)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Infantile Colic; Gastroesophageal Reflux (GER); Functional Constipation; Functional Diarrhea; Dysbiosis
Keywords: BioAmicus Complete; probiotic; multistrain probiotic; infant; functional gastrointestinal symptoms; Infant Gastrointestinal Symptom Questionnaire; gut microbiome; stool microbiome
MeSH Terms: conditions — Colic; Gastroesophageal Reflux; Dysbiosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two-arm, single-center trial in infants 0-24 months comparing BioAmicus Complete plus usual care versus usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioAmicus Complete + Usual Care (Experimental): Participants receive BioAmicus Complete (multistrain probiotic) oral drops in addition to usual care for infant functional GI symptoms. Product is administered by caregivers per protocol/label for 42 days; adherence is recorded. No other probiotic products are permitted during the study. Concomitant medications and routine management are allowed at the investigator's discretion.
  Interventions: Dietary Supplement: BioAmicus Complete; Other: Usual Care (No Probiotic)
- Usual Care Alone (Active Comparator): Participants receive standard clinical management per local practice for infant functional gastrointestinal symptoms. No probiotic supplementation is provided (participants are asked to avoid other probiotic products during the study). Concomitant medications and supportive care may be used as clinically indicated at the investigator's discretion.
  Interventions: Other: Usual Care (No Probiotic)

INTERVENTIONS:
Dietary Supplement: BioAmicus Complete — Oral liquid probiotic (multistrain) administered by caregivers per protocol/label for 42 days to infants with functional GI symptoms. Given as drops by mouth; dosing and administration instructions per protocol. No other probiotic products allowed during the study. Concomitant medications and routine management may be used as clinically indicated. Adherence is recorded; lot/batch number captured.
  Other Names: Multistrain Probiotic (BioAmicus Complete)
  Arms: BioAmicus Complete + Usual Care
Other: Usual Care (No Probiotic) — Standard clinical management for infant functional gastrointestinal symptoms per local practice. No probiotic supplementation is provided during the study period. Participants follow the same visit and assessment schedule as the intervention arm. Concomitant medications and supportive care may be used as clinically indicated.
  Other Names: Standard care; Routine clinical management

SUMMARY:
Infants often experience functional gastrointestinal symptoms (e.g., colic, excessive gas, regurgitation, constipation, or loose stools) that distress families and may reflect an imbalance of the gut microbiome. This study evaluates whether the multistrain probiotic BioAmicus Complete can improve caregiver-reported gastrointestinal symptoms in infants 0-24 months and is safe for use in this population.

The primary assessment is the change in the Infant Gastrointestinal Symptom Questionnaire (IGSQ) total score from the start to the end of the study period. Secondary assessments include symptom domains (colic/regurgitation, stool frequency and consistency), caregiver quality of life, growth parameters (weight and length), health care utilization and antibiotic exposure, and overall safety/tolerability (adverse events and serious adverse events). Stool samples will be analyzed to explore changes in the gut microbiome.

DETAILED DESCRIPTION:
caregiver burden and health care visits. Modulating the developing gut microbiome with probiotics may alleviate these symptoms. BioAmicus Complete is a multistrain probiotic designed to support a healthy intestinal microbiota; systematic clinical evaluation is warranted to determine its efficacy and safety in infants.

Objectives:

Primary: Determine whether BioAmicus Complete improves overall gastrointestinal symptoms versus usual care, measured by change in IGSQ total score between baseline and study end.

Exploratory (microbiome): Characterize changes in stool microbiome composition and diversity across the study period.

Secondary: Compare groups on symptom domain scores (e.g., colic, regurgitation, stooling patterns), caregiver burden/quality of life, health care utilization and antibiotic exposure, growth parameters, and safety outcomes (adverse events, serious adverse events, and product-related events).

Significance: Findings will inform whether BioAmicus Complete can be recommended as an adjunct to routine care for infant functional gastrointestinal symptoms and will provide preliminary insights into microbiome changes associated with symptom improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-24 months at enrollment.
* Infant has clinician-assessed functional gastrointestinal symptoms (e.g., colic/irritability, regurgitation, constipation, loose stools), judged suitable for study participation.
* Parent or legal guardian provides written informed consent and agrees to comply with study procedures (questionnaires/diaries and sample collection, if applicable).
* Caregivers agree to avoid other probiotic products during the study period, except as directed by the study team.

Exclusion Criteria:

* Major congenital gastrointestinal anomalies or known chronic gastrointestinal diseases requiring ongoing prescription therapy (e.g., Hirschsprung disease, inflammatory bowel disease, short-bowel syndrome).
* Clinically unstable condition or severe/critical illness that could interfere with participation or safety in the opinion of the investigator.
* Known or suspected primary or secondary immunodeficiency, or current immunosuppressive therapy.
* History of severe allergy or hypersensitivity to components of the investigational product.
* Recent use of systemic antibiotics within 14 days prior to baseline, or use of probiotic supplements within 14 days prior to baseline (per protocol).
* Participation in another interventional clinical trial within 30 days prior to enrollment or during the study.
* Any condition that, in the investigator's judgment, would make the participant unsuitable for the study or confound outcome assessments.

Ages: 0 Days to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Infant Gastrointestinal Symptom Questionnaire (IGSQ) Total Score at Day 42 | Baseline to Day 42
  IGSQ is a 13-item, caregiver-reported questionnaire (total score 13-65; higher scores indicate worse symptoms). Change is calculated as Day 42 minus baseline; a negative change indicates improvement
Stool Microbiome - Change in Alpha Diversity (Shannon, Chao1) | Baseline to Day 42
  16S rRNA gene sequencing of stool at baseline and Day 42; alpha diversity indices computed and change analyzed within and between groups.

SECONDARY OUTCOMES:
Change in Stool Frequency Based on Infant & Toddler GI Symptom Questionnaire from Baseline to Day 42 | Baseline to Day 42
  Stool frequency is assessed. Responses range from 1 (≤2 times/week) to 5 (>3 times/day). Higher scores indicate more frequent bowel movements (diarrhea tendency), while lower scores indicate infrequent stools (constipation). Improvement is defined as movement toward the normal category (1 bowel movement/day).
Change in Stool Consistency Using the Brussels Infant and Toddler Stool Scale (BITSS) from Baseline to Day 42 | Up to Day 42
  Stool consistency is assessed using the Brussels Infant and Toddler Stool Scale (BITSS), with five categories: 1 = watery, 2 = soft, 3 = formed, 4 = hard, 5 = inconsistent. Category 3 (formed) is considered normal. Scores below 3 represent looser stools (diarrhea tendency), while scores above 3 represent harder stools (constipation tendency). Improvement is defined as a ≥1-category change toward formed stool.
Stool Microbiome - Between-Group Difference in Beta Diversity (PERMANOVA) | Day 42
  Bray-Curtis and UniFrac distances used to assess community differences between groups; hypothesis testing via PERMANOVA.
Change in Frequency of Regurgitation and Vomiting Episodes from Baseline to Day 42 | Baseline to Day 42
  Regurgitation and vomiting are assessed using Questions. Frequency is reported on a 7-point ordinal scale (0 = never to 6 = >5 times/day). Higher scores indicate more frequent regurgitation/vomiting (worse outcome). Improvement is defined as a reduction of ≥1 category on the frequency scale.
Change in Colic Symptoms Based on Infant & Toddler GI Symptom Questionnaire from Baseline to Day 42 | Baseline to Day 42
  Colic is assessed, based on Wessel's criteria (≥3 hours/day, ≥3 days/week, for ≥3 weeks). Responses are scored on a binary scale (Yes/No). Presence of colic is considered a positive outcome at baseline. Improvement is defined as resolution of criteria (reduction below threshold)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial and Bioequivalence Center, Haiphong, Hai Phong, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcomes will be shared. Datasets will include: baseline characteristics; IGSQ item and total scores; caregiver diary data (stool frequency/form, regurgitation/vomiting counts, crying/irritability duration); growth parameters; concomitant medications; protocol deviations; and safety data (TEAEs/SAEs, relatedness, severity). For microbiome analyses, processed data (e.g., feature/ASV tables, relative abundance matrices, and diversity indices) will be shared; raw sequencing reads may be available on justified request. A data dictionary and variable codebook will accompany the IPD.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting materials will become available ~6 months after publication of the primary results and will remain available for 36 months thereafter. Earlier access may be granted for bona fide regulatory or public health needs. Extensions beyond 36 months will be considered upon reasonable request.
Access Criteria: Access is available to qualified researchers with a methodologically sound proposal and, where applicable, IRB/ethics approval or waiver. Submit requests to the study contacts listed in this record, including a brief proposal and analysis plan. Approved requestors must sign a Data Use Agreement; data will be provided via secure transfer. Data may be used only for the approved objectives; re-identification is prohibited; citation of the original study is required; data must be destroyed or returned at the end of the access period.